CLINICAL TRIAL: NCT01880385
Title: Efficacy & Safety of Bevacizumab as Neoadjuvant Treatment in Patients With Locally Advanced Inflammatory Breast Cancer, a Pilot Study.
Brief Title: Efficacy and Safety of Bevacizumab in the Neodjuvant Treatment of Inflammatory Breast Cancer
Acronym: Beva
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Association Tunisienne de lutte Contre le Cancer (Other)
Collaborators: Hoffmann-La Roche (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25168
Record Dates: First submitted 2011-05-25; First posted 2013-06-19 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Inflammatory Breast Cancer
Keywords: bevacizumab; inflammatory breast cancer; non metastatic; Avastin
MeSH Terms: conditions — Inflammatory Breast Neoplasms | interventions — Bevacizumab; Cyclophosphamide; Epirubicin; Fluorouracil; Docetaxel; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bevacizumab, inflammatory breast cancer (Experimental): Neoadjuvant therapy associating bevacizumab, cyclophosphamide, fluorouracil and epirubicin hydrochloride q3w, 4 cycles Adjuvant therapy by docetaxel q3w, 4 cycles +/- trastuzumab q3w, 18 cycles if tumors overexpress HER2
  Interventions: Biological: Bevacizumab; Drug: Cyclophosphamide; Drug: epirubicin hydrochloride; Drug: fluorouracil; Drug: Docetaxel; Biological: Trastuzumab

INTERVENTIONS:
Biological: Bevacizumab — During neoadjuvant phase: 15 mg/kg, d1 q3w, 4 cycles
  Other Names: Avastin
Drug: Cyclophosphamide — Neoadjuvant: 500 mg/m2 d1 q3w, 4 cycles
Drug: epirubicin hydrochloride — Neoadjuvant: 100 mg/m2, d1 q3w, 4 cycles
Drug: fluorouracil — Neoadjuvant: 500 mg/m2, d1 q3w, 4 cycles
Drug: Docetaxel — Adjuvant: 100 mg/m2 q3w, 4 cycles
Biological: Trastuzumab — Adjuvant: 8 mg/kg d1 in the 1st cycle then 6 mg/kg for d1 q3w, 17 cycles if tumor overexpress HER2

SUMMARY:
Multi-center, non randomised, open label, non controlled pilot study. Evaluating the treatment of bevacizumab in association with pre-operative chemotherapy, followed by surgery, adjuvant chemotherapy and radiotherapy in Patients with inflammatory breast cancer.

DETAILED DESCRIPTION:
Pilot study evaluating the safety and efficacy of adding Bevacizumab to neoadjuvant chemotherapy in patients presenting non metastatic inflammatory breast cancer (IBC). Patients will receive 4 cycles of chemotherapy FEC100 associating Fluorouracil (500 mg/m2), Epirubicin (100 mg/m2), Cyclophosphamide (500 mg/m2) and Bevacizumab 15 mg/kg every at day 1 of ecah 21 days cycle for 4 cycles. Six weeks after the end of neoadjuvant chemotherapy, patients will undergo mastectomy and 4 cycles of Docetaxel (100 mg/m2)as adjuvant chemotherapy +/-Trastuzumab 8 mg/kg for the first cycle then 6mg/kg every 3 weeks for 17 cycles if tumor overexpress Human Epidermal Growth Factor Receptor 2 (HER2).

The primary objective of this study is to evaluate the safety and the efficacy, i.e. pathologic complete response (pCR) after 4 cycles of FEC100+Bevacizumab in IBC

ELIGIBILITY:
Inclusion Criteria:

* • Patients must have signed a written informed consent form prior to any study specific procedures,

  * Women,
  * 20 years or older,
  * Performance status < 2 (ECOG),
  * Histologically confirmed inflammatory breast cancer T4d any N,
  * hormonal Status known,
  * no metastases according to the last TNM classification,
  * adequate hematologic function :

    * absolute neutrophil count ≥ 1 500/mm3
    * Platelets ≥ 100 000/mm3
    * Hemoglobin ≥ 9 g/dL
  * adequate liver function :

    * ASAT and ALAT < à 3 ULN
    * Alkaline Phosphatase < 5 ULN
    * Total bilirubin < 1,5 ULN, o
  * adequate kidney function :

    * creatinine < 1,5 x normal or creatinine Clearance ≥ 50ml/min (according to the cockcroft and Gault formula)
    * Urine Dipstick for proteinuria < 2+ patients who have proteinuria ≥ 2 + on dipstick urinalysis at baseline should undergo a 24 hours urine collection and must demonstrate ≤ 1 g of protein in 24 hours,
  * adequate coagulation and cardiac function :

    * Prothrombin ratio ≥ 70 % and,
    * Prothrombin time ≤ 1,5 upper limit of normal (ULN) within 7 days prior to enrolment
    * Left Ventricular ejection fraction (LVEF) ≥ 55 %

Exclusion Criteria:

* Patients of childbearing potential with a positive pregnancy test (serum or urine) prior to enrollment
* Patients who are either not post-menopausal, or surgically sterile, not using "effective contraception" (the definition of "effective contraception" will be based on the judgment of the investigator)
* Patients who are pregnant or breastfeeding
* Patient considered socially or psychological unable to comply with the treatment and the required medial follow-up,
* Concurrent participation in another clinical trial or treatment with any other anticancer agent during the protocol specified period
* Patients unwilling or unable to sign and date an Ethics Committee (EC)/ Institutional Review Board (IRB)-approved patient informed consent form
* Patients unwilling or unable to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
* Non inflammatory breast cancer with lymphatic skin permeation, Metastases,
* Bilateral breast cancer
* Distant metastases (stage IV)
* History of another cancer other than adequately treated carcinoma in situ of the cervix uteri, basal or squamous cell skin cancer
* Prior anti tumor therapy (surgery, radiotherapy, chemotherapy, hormonal treatment and targeted therapy) except treatments given for carcinoma in situ of the cervix uteri, basal or squamous cell skin cancer
* History or evidence of inherited bleeding diathesis or coagulopathy,
* History of thrombotic disorders within the last 6 months prior to enrollment (i.e. cerebrovascular accident, transient ischemic attacks, subarachnoid hemorrhage),
* Uncontrolled hypertension (systolic > 150 mmHg and/or diastolic > 100 mmHg)with or without any anti-hypertensive medication ; patients with high initial blood pressure are eligible if entry criteria are met after initiation or adjustment of anti-hypertensive medication,
* Any of the following within 6 months prior to enrollment:

myocardial infarction, severe/unstable angina, or coronary/peripheral artery bypass graft surgery, clinically symptomatic and uncontrolled cardiovascular disease, or clinically significant cardiac arrhythmias (grade 3-4)

* Severe resting dyspnea due to complications or oxygen dependency,
* Diabetic patient treated with oral anti-diabetics or insulin with an underlying cardiopathy at ultrasound,
* Any other severe acute illness such as active uncontrolled infections that would preclude the safe administration of study therapy at the time of the enrolment
* Other severe underlying medical conditions, which could impair the ability to participate in the study
* Major surgery, significant traumatic injury within 28 days prior to study treatment start or anticipation of the need for major surgery during study treatment,
* Minor surgery, including insertion of an indwelling catheter, within 24 hours prior to the first bevacizumab infusion,
* Non-healing wound, active peptic ulcer or bone fracture,
* History of abdominal fistula, diagnosed with a trachea-oesophageal fistula or any grade 4 non gastro-intestinal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months of enrolment,

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-09 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
pathologic Complete Response (pCR) | 18 months
  Evaluation of the pathologic complete response (pCR) rate among patients treated by 4 cycles of FEC100 and bevacizumab

SECONDARY OUTCOMES:
Toxicity as assessed by CTCAE v3.0 | 3 and 5 years
  Evaluation of the safety of administering bevacizumab in the neoadjuvant setting, with particular attention on the incidence of grade 3/4 adverse events
Progression-free survival | 3 and 5 years
Overall survival | 3 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: amel mezlini, professor, Principal Investigator — Institut Salah Azaiz
Locations (1):
- Institut Salah Azaiz, Bab Saadoun, Tunis Governorate, Tunisia

REFERENCES:
- [Background] Wedam SB, Low JA, Yang SX, Chow CK, Choyke P, Danforth D, Hewitt SM, Berman A, Steinberg SM, Liewehr DJ, Plehn J, Doshi A, Thomasson D, McCarthy N, Koeppen H, Sherman M, Zujewski J, Camphausen K, Chen H, Swain SM. Antiangiogenic and antitumor effects of bevacizumab in patients with inflammatory and locally advanced breast cancer. J Clin Oncol. 2006 Feb 10;24(5):769-77. doi: 10.1200/JCO.2005.03.4645. Epub 2006 Jan 3. PMID 16391297